CLINICAL TRIAL: NCT02263287
Title: LESCOD: "A Single Center, Prospective Study Aimed at Validating a Clinical Scale, Screening for Symptoms of Lewy Body Disease in Patients Incipient Dementia of the Alzheimer's and/or Lewy Body Type"
Brief Title: LESCOD: "Lewy Body Screening in Cognitive Disorders"
Acronym: LESCOD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment problems
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC14_0007
Record Dates: First submitted 2014-07-22; First posted 2014-10-13 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Alzheimer Disease; Lewy Body Disease
Keywords: Alzheimer Disease; Lewy Body Disease
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alzheimer disease (AD) (Other): Patients with AD according to NINCDS-ADRDA (National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association) criteria Intervention: LeSCoD scale
  Interventions: Other: LeSCoD scale
- Dementia with Lewy Bodies (DLB) (Other): Patients with probable DLB according to McKeith criteria. Intervention: LeSCoD scale
  Interventions: Other: LeSCoD scale
- Probable AD and possible DLB (Other): Patients with clinical criteria for possible or probable AD and possible DLB Intervention: LeSCoD scale
  Interventions: Other: LeSCoD scale

INTERVENTIONS:
Other: LeSCoD scale — LeSCoD is a clinical scale

SUMMARY:
Dementia with Lewy body (DLB) is the second most common neurodegenerative dementia in autopsy series. However, DLB represents a small proportion of the clinical diagnoses in epidemiology registries. Indeed Alzheimer disease (AD) and DLB are often concomitant, they share many symptoms and only a small weight is given to non-motor symptoms in DLB diagnosis. DLB is at the end of a pathological spectrum overlapping with AD, explaining the poor diagnostic value of both diagnostic criteria. To date there is still a need for a tool able to discriminate patients with pure DLB from those expressing common signs with both AD and DLB and those with pure AD. The purpose of this study is to validate a semi quantitative scale designed to reflect the Lewy Bodies burden in patients with mild to moderate cognitive decline. The investigators hypothesized that the score obtained may differentiate between AD, DLB and patients fulfilling clinical criteria for both DLB an AD. This score could also be correlated with dopaminergic depletion assessed with [18F]fluorodopa PET/computed tomography and/or with potential biomarkers of ADD measured in cerebrospinal fluid. This clinical validation is a preliminary work preceding further studies correlating the LeSCoD score with functional imaging features, prognosis and therapeutic response. Thus, the expected outcomes involve an improvement in demented patients' care, as well as a better patient selection for further therapeutic studies

ELIGIBILITY:
Inclusion Criteria:

* Be a woman or a male >60 to < 90 years
* Have sufficient visual and auditory acuity
* Be able to speak, read, hear and understand french language
* Be covered by health care insurance
* Have a reliable help/partner/informant/caregiver
* Have a mild to severe cognitive decline based on MMSE (Mini-Mental State Examination) score ( From 18 to 26)
* Give oral agreement to the assessment of the LEsCoD scale during routine consultation
* Have performed neuropsychology tests and MRI respectively within 6 and 12 months

Exclusion Criteria:

* Has evidence of neurological or psychiatric disorder other than AD or DLB explaining cognitive decline
* Has received previously or currently neuroleptic treatment
* Has no reliable help/caregiver the day of the visit
* Refuses to give his/her oral agreement to the assessment of the LeSCoD scale
* Has presence on MRI of radiologic evidence of cerebrovascular disease (score Fazekas 2)

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Construct validity of the LeSCoD scale with a factorial analysis | Day 0 (during the inclusion visit)
  The study consists in one single mandatory visit and 2 optional visits. The clinical scale is performed during the inclusion visit which corresponds to a routine consultation scheduled at the memory clinic

SECONDARY OUTCOMES:
Diagnostic validity of the Lescod scale by measuring the sensitivity and the specificity | Day 0 (During the inclusion visit)
  The study consists in one single mandatory visit and 2 optional visits. The clinical scale is performed during the inclusion visit which corresponds to a routine consultation scheduled at the memory clinic
Intergroup variance will be used to assess the quality of the patient denomination | Day 0 (during the inclusion visit)
  The study consists in one single mandatory visit and 2 optional visits. The clinical scale is performed during the inclusion visit which corresponds to a routine consultation scheduled at the memory clinic
Concurrent validity will be assessed by the measurement of the striatal dopaminergic depletion and its correlation with the Lescod score | Day 0 (during the inclusion visit)
  The study consists in one single mandatory visit and 2 optional visits. The clinical scale is performed during the inclusion visit which corresponds to a routine consultation scheduled at the memory clinic

CONTACTS AND LOCATIONS:
Overall Officials: Sarah EVAIN, Doctor, Study Chair — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France